CLINICAL TRIAL: NCT02218229
Title: The Effect of Extracorporeal Shock Wave Therapy on Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-102-05-122
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: shock wave; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shock waves (Experimental): Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs). Different studies and clinical experiments have demonstrated the efficacy of shock waves in the treatment of musculoskeletal system such as chronic tendinopathies or hypertrophic pseudoarthrosis.
  Interventions: Device: Shock wave
- Night splint (No Intervention): The wrist night splint was firmly fixed in a neutral position to immobilize the affected wrist. Patients were ordered to wear the splint while resting at night and at least 8 hours per day during the period of study

INTERVENTIONS:
Device: Shock wave — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs). Different studies and clinical experiments have demonstrated the efficacy of shock waves in the treatment of musculoskeletal system such as chronic tendinopathies or hypertrophic pseudoarthrosis
  Other Names: E-SWT, Elettronica Pagani, Italy
  Arms: Shock waves

SUMMARY:
The shock wave is a new and potential intervention for the reinnervation of peripheral nerve. The purpose of this study was to assess the effect of extracorporeal shock wave therapy on carpal tunnel syndrome.

DETAILED DESCRIPTION:
Recently, many studies show the potential effect of shock wave for the reinnervation for peripheral neuropathy in the animal mode. Only one study reveal the potential benefit of shock wave in patients with carpal tunnel syndrome. Althouh its expressive finding, the number of cases is relatively too small to make a conclusive remark. Large and well-designed study would expand the new field.

ELIGIBILITY:
Inclusion Criteria:

Outpatient subjects who had typical symptoms and signs of CTS, such as positive Tinel's sign or Phalen's test and numbness/tingling in at least two of the first, second, and third digits and were all confirmed by electrophysiological study, were considered and enrolled.

Exclusion Criteria:

The patients who had conditions mimicking CTS, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previous wrist surgery or steroid injection for CTS, were all excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on1st, 2nd, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 1st, 2nd, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th,12th and 16th weeks after treatment.
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline in cross-sectional area of the median nerve on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment.
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline in conduction velocity, ampliture of median nerve on 1st, 2nd, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th,12th and 16th weeks after treatment.
  The antidromic sensory nerve conduction velocityof the median nerve was performed on all subjects according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA). The median nerve was stimulated at the wrist between the palmar longus and flexor carpal radialis tendon at a distance of approximately 14 cm from the active electrode.
Change from baseline in finger pinch on 1st, 2nd, 4th, 8th, 12th and 16th weeks after treatment. | Pre-treatment, 1st, 2nd, 4th, 8th,12th and 16th weeks after treatment.
  The finger pinch strength was measured using Jamar dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Tri-Service General Hospital, School of Medicine, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, School of Medicine, National Defense Medical Center, Taipei, Neihu, Taiwan

REFERENCES:
- [Background] Stevens JC, Sun S, Beard CM, O'Fallon WM, Kurland LT. Carpal tunnel syndrome in Rochester, Minnesota, 1961 to 1980. Neurology. 1988 Jan;38(1):134-8. doi: 10.1212/wnl.38.1.134. PMID 3336444
- [Background] Orhan Z, Alper M, Akman Y, Yavuz O, Yalciner A. An experimental study on the application of extracorporeal shock waves in the treatment of tendon injuries: preliminary report. J Orthop Sci. 2001;6(6):566-70. doi: 10.1007/s007760100013. PMID 11793180
- [Background] Ohtori S, Inoue G, Mannoji C, Saisu T, Takahashi K, Mitsuhashi S, Wada Y, Takahashi K, Yamagata M, Moriya H. Shock wave application to rat skin induces degeneration and reinnervation of sensory nerve fibres. Neurosci Lett. 2001 Nov 23;315(1-2):57-60. doi: 10.1016/s0304-3940(01)02320-5. PMID 11711214
- [Background] Wu YH, Lun JJ, Chen WS, Chong FC. The electrophysiological and functional effect of shock wave on peripheral nerves. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:2369-72. doi: 10.1109/IEMBS.2007.4352803. PMID 18002469
- [Background] Romeo P, d'Agostino MC, Lazzerini A, Sansone VC. Extracorporeal shock wave therapy in pillar pain after carpal tunnel release: a preliminary study. Ultrasound Med Biol. 2011 Oct;37(10):1603-8. doi: 10.1016/j.ultrasmedbio.2011.07.002. Epub 2011 Aug 19. PMID 21856074